CLINICAL TRIAL: NCT03743701
Title: A Prospective Comparative Study to Improve Preoperative Ultrasound Diagnosis of Rectal Fistulas in the Formation of Topical Diagnosis Using B-mode and Three-dimensional Image Reconstruction.
Brief Title: Endorectal Three-dimensional Ultrasound in the Diagnosis of Cryptogenic Fistulas of the Rectum.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: State Scientific Centre of Coloproctology, Russian Federation (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 82
Record Dates: First submitted 2018-11-08; First posted 2018-11-16 (Actual); Last update posted 2018-11-16 (Actual); Status verified 2018-11

CONDITIONS: Anal Fistula
MeSH Terms: conditions — Rectal Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transrectal ultrasound in В-mode (Active Comparator)
  Interventions: Diagnostic Test: The method of transrectal ultrasound in В-mode
- Transrectal ultrasound examination using three-di (Experimental)
  Interventions: Diagnostic Test: The method of transrectal ultrasound examination using three-dimensional image reconstruction.

INTERVENTIONS:
Diagnostic Test: The method of transrectal ultrasound in В-mode — A linear transrectal ultrasonic sensor with a frequency of 9 MHz is inserted into the rectum lumen to a depth of 10 cm from the edge of the anus. In real time, the rectal wall and anatomical structures of the anal canal are evaluated using linear sections. The localization of the internal fistula opening, the course of the fistula relative to the fibers of the external sphincter and the presence or absence of cellular and wall plug is determined.
  Arms: Transrectal ultrasound in В-mode
Diagnostic Test: The method of transrectal ultrasound examination using three-dimensional image reconstruction. — A mechanical circular transrectal ultrasonic sensor with a frequency of 13 MHz is inserted into the rectum lumen to a depth of 10 cm from the edge of the anus. Within 30 seconds with a scan interval of 2 mm with a length of 10 cm, a circular recording of the anatomical structures of the rectum, surrounding tissue and anal canal takes place, obtaining an array of images in the form of a cube. The study was completed. After, at a convenient time for the researcher is working with a three-dimensional array of images. The resulting cube can be rotated 360 degrees in a circle of its axis, work with the sagittal, frontal and axial plane. To obtain a more visual representation of the exact localization of the internal fistula orifice, the course of the fistula relative to the fibers of the outer sphincter and to design volumetric cellular and wall plug.
  Arms: Transrectal ultrasound examination using three-di

SUMMARY:
Prospective comparative parallel ultrasound diagnostic transrectal study in the diagnosis of cryptogenic fistulas of the rectum

DETAILED DESCRIPTION:
It is planned to investigate 150 patients with cryptogenic fistulas. Patients will be divided into two groups: complete and incomplete internal fistulas of the rectum. Patients of the first group will undergo preoperative examination in the framework of transrectal ultrasound in B-mode, three-dimensional reconstruction of the image with a contrast of the fistula course with a solution of 1.5% hydrogen peroxide. Patients with incomplete internal fistulas of the rectum will also undergo transrectal ultrasound examination in B-mode and with three-dimensional image reconstruction. The results obtained in the two groups will be compared with the intraoperative revision.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with "fistula of the rectum"
* Patients diagnosed with cryptogenic fistulas
* Patients who have signed informed consent

Exclusion Criteria:

* Patients with perianal complications of Crohn's disease
* Рatients with post-traumatic fistulas
* Рatients with fistulas, drain pararectal cysts
* Рatients with anal fissures, complicated by rectal fistula
* Рatients who refused to participate in the study of their own free will

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 years and older
Enrollment: 150 (Estimated)
Dates: Start 2017-12-30 (Actual); Primary Completion 2020-08-31 (Estimated); Study Completion 2020-08-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 14 days
  Sensitivity in the diagnosis of cryptogenic fistulas of the rectum

CONTACTS AND LOCATIONS:
Locations (1):
- State Sceintific Centtre of Coloproctology, Moscow, Russia